CLINICAL TRIAL: NCT07197801
Title: Evaluation of a Peer Recovery Support Program Adapted to Target Retention in Clinic-based Medication for Opioid Use Disorder Treatment
Acronym: PEERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: UConn Health (Other)
Responsible Party: Principal Investigator, Melissa Poulsen, Associate Professor, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R33DA059880-02 (NIH)
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder
Keywords: Medication for opioid use disorder; Peer recovery support
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Study participants will receive the standard care - medication treatment for opioid use disorder
- Standard Care + Peer Recovery Support (Experimental): In addition to standard care (medication treatment for opioid use disorder), study participants will receive support provided by a peer recovery support specialist
  Interventions: Behavioral: Peer recovery support to enhance patient engagement in medication for opioid use disorder treatment

INTERVENTIONS:
Behavioral: Peer recovery support to enhance patient engagement in medication for opioid use disorder treatment — The intervention adds a peer recovery support (PRS) program to standard outpatient medication for opioid use disorder treatment and medical care. The PRS program will entail meeting one-on-one with a peer recovery specialist over a 6-month period, who will utilize their lived experience with substance use and recovery to provide emotional, informational, instrumental, and aﬃliational support to participants.
  Arms: Standard Care + Peer Recovery Support

SUMMARY:
The goal of this clinical trial is to learn if receiving peer recovery support (support services provided by trained "peers" with lived experience of addiction and recovery) improves retention in medication treatment among people with opioid use disorder. The main question it aims to answer is: does peer recovery support improve retention in medication treatment for opioid use disorder?

Researchers will compare two groups: (1) standard care combined with a peer recovery support program, and (2) standard care alone, to see if peer recovery support works to improve retention in medication treatment for opioid use disorder.

Participants will: visit clinics as they normally would to receive standard care (medication treatment for opioid use disorder); complete two questionnaires - one when they start treatment and one 6 months later; and agree to let researchers use information from their medical record. Participants in group 1 will also be invited to meet with a peer recovery support specialist for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years of age
* Initiated medication for opioid use disorder treatment in past 45 days in a Geisinger outpatient clinic
* Willing and able to give informed consent

Exclusion Criteria:

* Received medication for opioid use disorder treatment at a Geisinger outpatient clinic in the 90-day period prior to the treatment initiation date
* Not proficient in English

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
6-month treatment retention | 180 days from initiation of medication treatment for opioid use disorder
  Data will come from the electronic health records. Retention will be defined as a participant not having a lapse in days' supply of medication for opioid use disorder treatment (buprenorphine, buprenorphine-naloxone, or naltrexone) within the 6-month follow-up period that is greater than 30 days.
Length of time in treatment | 180 days from initiation of medication treatment for opioid use disorder
  Data will come from the electronic health records. Length of time in treatment will be determined by summing days' supply of consecutive orders for medications for opioid use disorder treatment(buprenorphine, buprenorphine- naloxone, or naltrexone). Treatment will be considered ended if a participant has a gap in supply of more than 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Poulsen, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A dataset from the randomized controlled trial (RCT) of U.S. adult patients initiating medication for opioid use disorder treatment will be shared. The data will be obtained from electronic health records (EHRs) and two assessments completed by study participants at baseline and 6-months follow-up. Data elements include each patients' study group assignment (standard care (SC) or SC plus the peer recovery support program), study outcomes, demographic and clinical covariates, and potential mediating and moderating variables. A second dataset from the subset of individuals randomized to SC+PRS will be shared. This data will come from a combination of EHRs, study logs, and assessments completed by patients. Data includes variables pertaining to patient's degree of engagement and satisfaction with the PRS program.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be released when study results are published, or at the end of the granting period, whichever comes first. Data will be permanently archived.
Access Criteria: De-identified datasets and meta-data will be available to access via the National Addiction & HIV Data Archive Program (NAHDAP) repository. Accessing data will require user registration and agreement to the data repository's terms of use, which require users to make no attempt to identify human subjects, cite the data/DOI, and not redistribute the data without NAHDAP written permission.